CLINICAL TRIAL: NCT03961945
Title: Minimally Invasive Molecular Approaches for the Diagnosis of Barrett's Esophagus and Esophageal Adenocarcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-002629; R01CA241164 (NIH); NCI-2021-14395 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-05-15; First posted 2019-05-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Barrett Esophagus; Esophageal Adenocarcinoma
Keywords: Barrett's Esophagus; Gastroesophageal Reflux; Reflux; Esophageal Cancer; Esophageal Adenocarcinoma
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus; Gastroesophageal Reflux; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Screening Population (Other): Those that have gastroesophageal reflux or other risk factors for Barrett's Esophagus will be contacted and if agreeable undergo sponge capsule procedure and fill out questionnaires.
  Interventions: Device: Sponge Capsule
- Upper endoscopy - Barrett's Esophagus (Other): Those that have a diagnosis of Barrett's Esophagus and are scheduled for an upper endoscopy will be approached and if agreeable undergo sponge capsule procedure as well as endoscopic biopsies and brushings of the esophagus.
  Interventions: Device: Sponge Capsule
- Upper endoscopy - No Barrett's Esophagus (Other): Those that have no known Barrett's Esophagus and are scheduled for an upper endoscopy will be approached and if agreeable undergo sponge capsule procedure as well as endoscopic biopsies and brushings of the esophagus.
  Interventions: Device: Sponge Capsule

INTERVENTIONS:
Device: Sponge Capsule — Subjects will swallow sponge capsule and esophageal cells will be collected on deployed sponge.
  Other Names: EsophaCap; Cytosponge

SUMMARY:
This study will evaluate if the sponge capsule device can accurately detect the presence of Barrett's Esophagus and prevalent dysplasia/adenocarcinoma detection, in a screening population, with and without chronic gastroesophageal reflux disease.

DETAILED DESCRIPTION:
The sponge on a string (SOS) device will be safely administered by a non-physician such as a nurse. Novel discriminant methylated DNA markers will be assayed on esophageal cytology specimens obtained from the SOS device to enable detection in Barrett's Esophagus and prevalent dysplasia/adenocarcinoma detection.

ELIGIBILITY:
Inclusion Criteria Aim1:

* Male and female ages 50-85
* Patients who have three or more risk factors for Barrett's Esophagus.
* Gastroesophageal reflux disease defined by:

  * Diagnosis
  * Use of one of the following drugs >= 3 months over the last 5 years: omeprazole, esomeprazole, pantoprazole, rabeprazole, dexlansoprazole, lansoprazole, ranitidine, famotidine, cimetidine
  * prior endoscopic diagnosis of erosive esophagitis
* Body mass index (BMI) >= 30

Exclusion Criteria Aim1 and Aim 3:

* Previous history of:

  * esophageal adenocarcinoma/cancer
  * esophageal squamous carcinoma
  * endoscopic ablation for Barrett's esophagus
  * esophageal squamous dysplasia
* Current treatment with oral anticoagulation including Warfarin, Coumadin
* History of cirrhosis
* History of esophageal/gastric varices
* History of Barrett's esophagus
* Prior endoscopy in the last 5 years

Inclusion criteria Aim 2 and Aim 3:

* Subjects with known or suspected BE (cases).

  * Patient between the ages 18 - 90.
  * Patients with a BE segment ≥ 1cm in maximal extent endoscopically or suspected BE in medical record.
  * Histology showing evidence of intestinal metaplasia with or without presence of dysplasia or suspected BE in medical record.
  * Undergoing clinically indicated endoscopy.
* Subjects without known history of BE (controls).

  * Undergoing clinically indicated diagnostic endoscopy.

Exclusion criteria Aim 2:

* Subjects with known BE.

  * Patients with prior history of ablation (photodynamic therapy, radiofrequency ablation, cryotherapy, argon plasma coagulation). Patients with history of endoscopic mucosal resection (EMR)/endoscopic submucosal dissection (ESD) alone will not be excluded.
  * Patients with history of esophageal resection for esophageal carcinoma.
* For subjects with or without known evidence of BE (on history or review of medical records):

  * Pregnant or lactating females.
  * Patients who are unable to consent.
  * Patients with current history of uninvestigated dysphagia (this does not apply to the brushings/biopsies only portion of the study).
  * History of eosinophilic esophagitis, achalasia.
  * Patients on oral anticoagulation including Coumadin, Warfarin (this does not apply to the brushings/biopsies only portion of the study).
  * Patients on antiplatelet agents including Clopidogrel, unless discontinued for three to five days prior to the sponge procedure.
  * Patients on oral thrombin inhibitors including Dabigatran and oral factor Xa inhibitors such as rivaroxaban, apixaban and edoxaban, unless discontinued for three to five days prior to the sponge procedure.
  * Patients with history of known esophageal or gastric varices or cirrhosis.
  * Patients with history of surgical esophageal resection for esophageal carcinoma.
  * Patients with congenital or acquired bleeding diatheses.
  * Patients with a history of esophageal squamous dysplasia.
  * Patient has known carcinoma of the foregut (pancreatic, bile duct, ampullary, stomach, or duodenum) within 5 years prior to study enrollment.
  * Patient has received chemotherapy class drugs or radiation to treat mediastinal or esophageal cancer.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1550 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2030-07-30 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
Aim 1 - Screening Population | 5 years
  To measure the positive and negative predictive value of the sponge capsule Barrett's esophagus test in a screening population.
Aim 2 - Case/Control Population BE Detection | 5 years
  Compare the sensitivity and specificity of a predetermined BE prediction algorithm for those with and without GERD and assess the influence of other covariates (age, sex, ever smoking, ethnicity and BMI) on this algorithm.
Aim 3 - Dysplasia Detection Sensitivity and Specificity | 5 years
  Measure the sensitivity and specificity of a predetermined MDM panel assayed on SOS specimens from BE patients identified in Aims 1 and 2, for the detection of HGD /EAC, using surveillance histology as the criterion standard.

SECONDARY OUTCOMES:
Aim 1 - Screening Population Predictive Value | 5 years
  Compare positive predictive value and negative predictive value of the sponge capsule Barrett's Esophagus test between those with and without chronic GERD.
Aim 1 - Screening Population Safety and Tolerability of sponge capsule procedure | 5 years
  Safety and tolerability of the sponge capsule device in a screening population as measured by a Tolerability Questionnaire with sponge capsule procedure. Participants will rate their tolerability by rating questions using a scale of 0-10 (0 is none and 10 is severe or 0 is good and 10 is not good).
Aim 2 - Case/Control Population Sensitivity and Specificity | 5 years
  Validate specificity and sensitivity cut offs of a BE prediction algorithm in an independent patient cohort
Aim 3 - Dysplasia Detection Rate of Missed Dysplasia | 5 years
  Measure diagnostic uncertainty bias in the criterion standard, specifically, the rate of dysplasia missed by surveillance histology

CONTACTS AND LOCATIONS:
Overall Officials: Prasad G. Iyer, M.D., Principal Investigator — Mayo Clinic
Locations (9):
- United States (9):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Mayo Clinic Health Systems - Austin, Austin, Minnesota
  - Mayo Clinic Health Systems - Mankato, Mankato, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Northwell Health, New Hyde Park, New York
  - Baylor Scott & White Research Institute, Dallas, Texas
  - Mayo Clinic Health System-Eau Claire, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials